CLINICAL TRIAL: NCT03044613
Title: Phase IB Trial of Induction Nivolumab or Nivolumab/Relatlimab Prior to Concurrent Chemoradiation in Patients With Operable Stage II/III Esophageal/ Gastroesophageal Junction Cancer
Brief Title: Nivolumab +/- Relatlimab Prior to Chemoradiation With II/III Gastro/Esophageal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1714; IRB00122689 (Other: JHMIRB)
Record Dates: First submitted 2017-01-25; First posted 2017-02-07 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer; Esophageal Cancer; GastroEsophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Nivolumab; relatlimab; Carboplatin; Paclitaxel; Taxes; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Nivolumab 240mg administered IV over 30 minutes every 2 weeks for 2 cycles and then standard of care chemoradiation (weekly carboplatin/paclitaxel and concurrent radiation
  Interventions: Drug: Nivolumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation
- Arm B (Experimental): Nivolumab 240mg administered IV over 30 minutes followed by relatlimab 80mg administered IV over 60 minutes on Day 1 every 2 weeks for 2 cycles and then standard of care chemoradiation (weekly carboplatin/paclitaxel and concurrent radiation).
  Interventions: Drug: Nivolumab; Drug: Relatlimab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation

INTERVENTIONS:
Drug: Nivolumab — 240mg or 1 mg/kg administered IV
  Other Names: Opdivo
Drug: Relatlimab — 80mg administered IV
  Other Names: BMS-986016; Anti-LAG3
  Arms: Arm B
Drug: Carboplatin — standard care dose
  Other Names: Paraplat; Paraplatin; Blastocarb; Carboplat; Carbosin; Carbosol; Carbotec; Displata; Ercar; Nealorin; Novoplatinum; Paraplatin AQ; Paraplatine; Platinwas
Drug: Paclitaxel — standard care dose
  Other Names: Taxol, Anzatax, Asotax, Bristaxol, Praxel, Taxol Konzentrat
Radiation: Radiation — standard care dose

SUMMARY:
Anti-PD-1 (nivolumab) or Anti-PD1/Anti LAG-3- (relaltimab) administration in the pre-operative setting with chemoradiation will be safe and feasible in patients with resectable distal esophageal/gastroesophageal junction cancer and will change cellular and molecular characteristics of the tumor microenvironment that will improve survival.

DETAILED DESCRIPTION:
This is a Phase IB study assessing the safety of 2 cycles of induction (Arm A) nivolumab or (Arm B) 2 cycles of induction nivolumab prior to concurrent chemoradiation plus nivolumab (Arm A) or nivolumab/relatlimab (Arm B) before surgical resection in operable stage II/III esophageal/gastroesophageal junction cancer.

Approximately 32 patients will be enrolled on study with 16 enrolled on Arm A and if no unexpected toxicities then an additional 16 patients will be enrolled on Arm B.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years old
* Histologically proven (squamous cell or adenocarcinoma) esophageal or gastro- esophageal junction cancer (core biopsy required).
* Stage II/III disease as per AJCC staging 7.0
* Baseline imaging with FDG-PET scan and endoscopic ultrasound within 28 days prior to registration
* ECOG performance status 0-1 (see Appendix B).
* Adequate oral intake/nutritional status without the need for enteral or parenteral feeding during chemoradiation or preoperative period
* Adequate organ function as follows:

  * Leukocytes ≥ 2,000/mm3
  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Creatinine ≤ 2.0 mg/dL
  * Bilirubin (total) within normal institutional limits (except subjects with Gilbert Syndrome who must have total bilirubin < 3.0 mg/dL)
  * AST(SGOT), ALT(SGPT), and alkaline phosphatase ≤ 2.5 times the upper limit of normal
  * PT such that international normalized ratio (INR) is ≤ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin and a PTT ≤ upper limit of normal
* Adequate cardiac function as defined by: no evidence of PR prolongation or AV block on baseline electrocardiogram (ECG).
* Radiation oncology consultation within 28 days to confirm that disease can be encompassed in the radiotherapy field and that normal tissue constraints can be met.
* Subjects must have adequate lung function to permit surgical resection determined by pre-enrollment pulmonary function tests to include DLCO as follows:

  * DLCO≥70% predicted OR DLCO<70% but ≥55% with a VO2 max ≥10L/min/kg (assessed by cardiopulmonary exercise testing) or 6 minute walk test ≥500 meters
  * Subjects with a DLCO<55% are excluded from this study.
  * Subjects must have a baseline O2 saturation by pulse oximetry that is ≥ 92% both at rest and while walking, off supplemental oxygen
* Esophagogastrectomies will be performed via a laparotomy and a right thoracotomy with en-bloc removal of perigastric, celiac, periesophageal and subcarinal lymph nodes. Esophagogastric reconstruction will be performed above the level of the azygo-caval junction using an EEA stapling device.
* Either a formalin fixed paraffin block or a minimum of ten 5-micron tissue section's (slides) of tumor biopsy sample must be available for biomarker evaluation from baseline and repeat EGD.
* The effects of nivolumab, on the developing human fetus are unknown. For this reason women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 5 months after the last dose of nivolumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Sexually active fertile men must use effective barrier birth control if their partners are WOCBP for 7 months after the last dose of nivolumab. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of registration.
* Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report AEs, understand the drug dosing schedule and use of medications to control AEs.
* (Relatlimab arm only) LVEF (Left Ventricular Ejection Fraction) assessment with documented LVEF ≥ 50% by either TTE or MUGA (TTE preferred test) within 6 months from first study drug administration

Exclusion Criteria:

* Patient has active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Esophageal tumors that are located in the mid esophagus or higher i.e. not involving distal esophagus or GE junction.
* Tumors whose proximal end are higher that the level of the carina
* Biopsy proven involvement of supraclavicular lymph nodes
* Tumors must not extend 5cm or more into the stomach
* Patient has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first dose. Inhaled or topical steroids and adrenal replacement steroid doses are permitted in the absence of active autoimmune disease.
* Subjects with previous malignancies (except non-melanoma skin cancers, in situ bladder, gastric, breast, colon or cervical cancers/dysplasia) are excluded unless a complete remission was achieved at least 1 years prior to study entry and no additional therapy (other than adjuvant hormonal therapy for breast cancer) is required or anticipated to be required during the study period.
* Subjects with brain metastasis are excluded from this study and all patients should have brain imaging (either MRI brain or CT brain with contrast) prior to enrollment.
* Subjects with a history of interstitial lung disease.
* Active systemic infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
* Known positive history or positive test for Human Immunodeficiency Virus or Acquired ImmunoDeficiency Syndrome (AIDS).
* History of allergy to study drug components.
* Women who are pregnant or nursing.
* WOBP and Men with female partners (WOCBP) that are not willing to use contraception.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-regulatory pathways).
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
* Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.
* (Relatlimab arm only) Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Subjects with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤1 x ULN. If TnT or TnI levels are > 1 to 2 × ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the BMS Medical Monitor or designee. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the BMS Medical Monitor or designee.
* (Relatlimab arm only) Participants must not have a history of myocarditis
* (Relatlimab arm only) Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
  * Uncontrolled angina within the 3 months prior to consent
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, poorly controlled atrial fibrillation, ventricular fibrillation, or torsades de pointes)
  * QTc prolongation > 480 msec
  * History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, , poorly controlled venous thrombosis etc.)
  * Cardiovascular disease-related requirement for daily supplemental oxygen
  * History of two or more MIs OR two or more coronary revascularization procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 100 days
  To investigate the safety of induction nivolumab or nivolumab/relatlimab administration prior to concurrent chemoradiation and nivolumab or nivolumab/relatlimab in subjects with resectable stage II/III gastro-esophageal junction cancer.

SECONDARY OUTCOMES:
Feasibility is assessed through the proportion of eligible patients who proceed to surgery without substantial delay (more than 60 days) due to treatment-related reasons | 12 weeks
  To investigate the feasibility of induction nivolumab or nivolumab/relatlimab prior to concurrent chemoradiation and nivolumab or nivolumab/relatlimab administration in subject's with stage II/III esophageal and gastro-esophageal junction cancer.
Pathological Complete Response Rate | 2 years
  To determine the pathological complete response rate in patients treated with induction checkpoint inhibition followed by chemo-radiation plus nivolumab prior to surgical resection
Approximate quantitation of infused nivolumab bound to PD-1 receptors on the surface of T cells in the peripheral blood and within the resected tumor and lymph node specimens | 2 years
  To explore the association between nivolumab +/-relatlimab exposure and selected pharmacodynamics markers in the peripheral blood and in the tumor microenvironment, including measurement of PD-1 receptor occupancy on tumor infiltrating lymphocytes.
Changes in Expression of Selected Immune Markers | 2 years
  To measure changes in expression of selected immune markers including changes in the quality and quantity of tumor infiltrating lymphocytes and the T effector to T-Reg ratio compared to baseline, in the blood, primary tumor tissue and draining lymph nodes
Overall Survival | 2 years
  To assess overall survival in patients receiving neoadjuvant checkpoint inhibitors.
Recurrence-Free Survival | 2 years
  To assess recurrence-free survival in patients receiving neoadjuvant checkpoint inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lam, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Alleghany Health Network, Pittsburgh, Pennsylvania
  - Baylor University/ Charles A. Sammons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] Lordick F, Ott K, Krause BJ, Weber WA, Becker K, Stein HJ, Lorenzen S, Schuster T, Wieder H, Herrmann K, Bredenkamp R, Hofler H, Fink U, Peschel C, Schwaiger M, Siewert JR. PET to assess early metabolic response and to guide treatment of adenocarcinoma of the oesophagogastric junction: the MUNICON phase II trial. Lancet Oncol. 2007 Sep;8(9):797-805. doi: 10.1016/S1470-2045(07)70244-9. PMID 17693134
- [Background] Moons LM, Kusters JG, Bultman E, Kuipers EJ, van Dekken H, Tra WM, Kleinjan A, Kwekkeboom J, van Vliet AH, Siersema PD. Barrett's oesophagus is characterized by a predominantly humoral inflammatory response. J Pathol. 2005 Nov;207(3):269-76. doi: 10.1002/path.1847. PMID 16177953
- [Background] Fitzgerald RC, Abdalla S, Onwuegbusi BA, Sirieix P, Saeed IT, Burnham WR, Farthing MJ. Inflammatory gradient in Barrett's oesophagus: implications for disease complications. Gut. 2002 Sep;51(3):316-22. doi: 10.1136/gut.51.3.316. PMID 12171950
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Llosa NJ, Cruise M, Tam A, Wicks EC, Hechenbleikner EM, Taube JM, Blosser RL, Fan H, Wang H, Luber BS, Zhang M, Papadopoulos N, Kinzler KW, Vogelstein B, Sears CL, Anders RA, Pardoll DM, Housseau F. The vigorous immune microenvironment of microsatellite instable colon cancer is balanced by multiple counter-inhibitory checkpoints. Cancer Discov. 2015 Jan;5(1):43-51. doi: 10.1158/2159-8290.CD-14-0863. Epub 2014 Oct 30. PMID 25358689
- [Background] Muro K, Chung HC, Shankaran V, Geva R, Catenacci D, Gupta S, Eder JP, Golan T, Le DT, Burtness B, McRee AJ, Lin CC, Pathiraja K, Lunceford J, Emancipator K, Juco J, Koshiji M, Bang YJ. Pembrolizumab for patients with PD-L1-positive advanced gastric cancer (KEYNOTE-012): a multicentre, open-label, phase 1b trial. Lancet Oncol. 2016 Jun;17(6):717-726. doi: 10.1016/S1470-2045(16)00175-3. Epub 2016 May 3. PMID 27157491
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Thompson ED, Zahurak M, Murphy A, Cornish T, Cuka N, Abdelfatah E, Yang S, Duncan M, Ahuja N, Taube JM, Anders RA, Kelly RJ. Patterns of PD-L1 expression and CD8 T cell infiltration in gastric adenocarcinomas and associated immune stroma. Gut. 2017 May;66(5):794-801. doi: 10.1136/gutjnl-2015-310839. Epub 2016 Jan 22. PMID 26801886
- [Background] Wu C, Zhu Y, Jiang J, Zhao J, Zhang XG, Xu N. Immunohistochemical localization of programmed death-1 ligand-1 (PD-L1) in gastric carcinoma and its clinical significance. Acta Histochem. 2006;108(1):19-24. doi: 10.1016/j.acthis.2006.01.003. Epub 2006 Mar 13. PMID 16530813
- [Background] Hou J, Yu Z, Xiang R, Li C, Wang L, Chen S, Li Q, Chen M, Wang L. Correlation between infiltration of FOXP3+ regulatory T cells and expression of B7-H1 in the tumor tissues of gastric cancer. Exp Mol Pathol. 2014 Jun;96(3):284-91. doi: 10.1016/j.yexmp.2014.03.005. Epub 2014 Mar 20. PMID 24657498
- [Background] Geng Y, Wang H, Lu C, Li Q, Xu B, Jiang J, Wu C. Expression of costimulatory molecules B7-H1, B7-H4 and Foxp3+ Tregs in gastric cancer and its clinical significance. Int J Clin Oncol. 2015 Apr;20(2):273-81. doi: 10.1007/s10147-014-0701-7. Epub 2014 May 9. PMID 24804867
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Background] Demaria S, Golden EB, Formenti SC. Role of Local Radiation Therapy in Cancer Immunotherapy. JAMA Oncol. 2015 Dec;1(9):1325-32. doi: 10.1001/jamaoncol.2015.2756. PMID 26270858
- [Background] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Rutkowski MR, Stephen TL, Svoronos N, Allegrezza MJ, Tesone AJ, Perales-Puchalt A, Brencicova E, Escovar-Fadul X, Nguyen JM, Cadungog MG, Zhang R, Salatino M, Tchou J, Rabinovich GA, Conejo-Garcia JR. Microbially driven TLR5-dependent signaling governs distal malignant progression through tumor-promoting inflammation. Cancer Cell. 2015 Jan 12;27(1):27-40. doi: 10.1016/j.ccell.2014.11.009. Epub 2014 Dec 18. PMID 25533336
- [Background] Goodman AL, Kallstrom G, Faith JJ, Reyes A, Moore A, Dantas G, Gordon JI. Extensive personal human gut microbiota culture collections characterized and manipulated in gnotobiotic mice. Proc Natl Acad Sci U S A. 2011 Apr 12;108(15):6252-7. doi: 10.1073/pnas.1102938108. Epub 2011 Mar 21. PMID 21436049
- [Derived] Kelly RJ, Landon BV, Zaidi AH, Singh D, Canzoniero JV, Balan A, Hales RK, Voong KR, Battafarano RJ, Jobe BA, Yang SC, Broderick S, Ha J, Marrone KA, Pereira G, Rao N, Borole A, Karaindrou K, Belcaid Z, White JR, Ke S, Amjad AI, Weksler B, Shin EJ, Thompson E, Smith KN, Pardoll DM, Hu C, Feliciano JL, Anagnostou V, Lam VK. Neoadjuvant nivolumab or nivolumab plus LAG-3 inhibitor relatlimab in resectable esophageal/gastroesophageal junction cancer: a phase Ib trial and ctDNA analyses. Nat Med. 2024 Apr;30(4):1023-1034. doi: 10.1038/s41591-024-02877-z. Epub 2024 Mar 19. PMID 38504015